CLINICAL TRIAL: NCT05599685
Title: A Non-interventional, Multicenter, Prospective stUdy to Record Treatment patteRns of nivOlumab+Ipilimumab+chemotheRapy Combination as First Line treAtment of Metastatic NSCLC in Routine Clinical Practice in Greece - the 'AURORA' Study
Brief Title: A Study of Nivolumab, Ipilimumab, and Chemotherapy in Participants With Non-small Cell Lung Cancer
Acronym: AURORA
Status: Recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-6PK
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non-small-cell lung cancer; NSCLC; nivolumab; ipilimumab; platinum-based chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants with metastatic NSCLC initiated on 1L treatment with NIVO/IPI/PBC

SUMMARY:
The purpose of this study is to describe the real-world patient and disease characteristics of metastatic non-small cell lung cancer (NSCLC) participants initiated on first-line (1L) treatment with nivolumab, ipilimumab, and platinum-based chemotherapy (NIVO/IPI/PBC), in the overall study population and the subpopulations per histological subtype of NSCLC and PD-L1 expression level.

ELIGIBILITY:
Inclusion Criteria:

* Participants with histologically- or cytologically-confirmed diagnosis of metastatic NSCLC (of any histological subtype) whose tumors have no sensitizing EGFR mutation or ALK translocation.
* Participants who have been initiated on 1L treatment with NIVO/IPI/PBC (nivolumab combined with ipilimumab and 2 cycles of PBC) as per the products' Summary of Product Characteristics (SmPC) prior to informed consent obtainment, and for whom the treatment regimen is ongoing and no more than one nivolumab infusion has been administered from treatment initiation to obtaining the signed informed consent.
* Participants for whom the decision to prescribe treatment with NIVO/IPI/PBC has been taken prior to their enrollment in the study and is clearly separated from the physician's decision to include the participant in the current study.

Exclusion Criteria:

* Participants with a current primary diagnosis of a cancer other than NSCLC that requires systemic or other treatment.
* Participants who have been treated with any prior systemic therapy in the metastatic setting of NSCLC.
* Participants who are currently receiving or are planned to receive treatment with any investigational drug/device/intervention or who have received any investigational product within 1 month or 5 half-lives of the investigational agent (whichever is longer) prior to NIVO/IPI/PBC therapy initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with metastatic non-small cell lung cancer initiated on first-line treatment with nivolumab, ipilimumab, and platinum-based chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-10-19 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Baseline participant and disease characteristics of interest in the overall study population and the subpopulations per NSCLC histological subtype and PD-L1 expression level | Baseline
Number of NIVO/IPI/PBC doses administered in the overall study population and the subpopulations per NSCLC histological subtype and PD-L1 expression level | Up to 157 weeks
Time interval between infusions in the overall study population and the subpopulations per NSCLC histological subtype and PD-L1 expression level | Up to 157 weeks
Rate of dose modifications in the overall study population and the subpopulations per NSCLC histological subtype and PD-L1 expression level | Up to 157 weeks
Rate of permanent treatment discontinuation in the overall study population and the subpopulations per NSCLC histological subtype and PD-L1 expression level | Up to 157 weeks
Frequencies of reasons for dose modifications/discontinuations in the overall study population and the subpopulations per NSCLC histological subtype and PD-L1 expression level | Up to 157 weeks
Cumulative dose of NIVO and IPI administered in the overall study population and the subpopulations per NSCLC histological subtype and PD-L1 expression level | Up to 157 weeks
Relative dose intensity (RDI) in the overall study population and the subpopulations per NSCLC histological subtype and PD-L1 expression level | Up to 157 weeks
  RDI (%) will be calculated as follows:
  For NIVO: [Cumulative dose (mg)/((Last Nivolumab dose date - Nivolumab Start dose date + 21) x 360/21)] x 100] For IPI: [Cumulative dose (mg)/((Last Ipilimumab dose date - Ipilimumab Start dose date + 21) x 360/21)] x 100]
Proportion of participants receiving ≥90% RDI of NIVO and IPI in the overall study population and the subpopulations per NSCLC histological subtype and PD-L1 expression level | Up to 157 weeks
Time from NIVO/IPI/PBC initiation until discontinuation due to any reason in the overall study population and the subpopulations per NSCLC histological subtype and PD-L1 expression level | Up to 157 weeks
Proportions of participants surviving at the landmark timepoints of 12, 24, and 36 months after NIVO/IPI/PBC initiation in the overall study population and the subpopulations per NSCLC histological subtype and PD-L1 expression level | 12, 24, and 36 months

SECONDARY OUTCOMES:
Proportions of participants who have not progressed or died from any cause at 12, 24, and 36 months after NIVO/IPI/PBC initiation in the overall study population and the subpopulations per NSCLC histological subtype and PD-L1 expression level | 12, 24, and 36 months
Proportions of participants with an investigator-assessed best overall response (BOR) of either a confirmed complete response (CR) or partial response (PR) after NIVO/IPI/PBC initiation in the overall population and the NSCLC and PD-L1 subpopulations | 12, 24, and 36 months
Proportions of participants with an investigator-assessed BOR of a confirmed CR, PR, or stable disease (Disease Control Rate (DCR)) after NIVO/IPI/PBC initiation in the overall study population and the NSCLC and PD-L1 subpopulations | 12, 24, and 36 months
Time from start of NIVO/IPI/PBC treatment to the first documented investigator-assessed response (CR or PR), among participants who achieved at least PR in the overall study population and the NSCLC and PD-L1 subpopulations | Up to 157 weeks
Time from first documented response to progression or death due to any cause in the absence of progression (Kaplan Meier DoR), among participants who achieved at least PR in the overall study population and the NSCLC and PD-L1 subpopulations | Up to 157 weeks
Types of next treatment planned to be administered for NSCLC after NIVO/IPI/PBC discontinuation in the overall study population and the subpopulations per NSCLC histological subtype and PD-L1 expression level | Up to 157 weeks
Frequencies of next treatment planned to be administered for NSCLC after NIVO/IPI/PBC discontinuation in the overall study population and the subpopulations per NSCLC histological subtype and PD-L1 expression level | Up to 157 weeks
Exposure-adjusted incidence rate (EAIR) of the following types of treatment-related AEs in the overall study population | Up to 157 weeks
  * Select irAEs: Immune-related pneumonitis, immune-related colitis, immune-related hepatitis, immune-related nephritis and renal dysfunction, immune-related endocrinopathies (hyperthyroidism, hypothyroidism, adrenal insufficiency, hypophysitis, diabetes mellitus and diabetic ketoacidosis), and immune-related skin adverse reactions (rash, Stevens-Johnson syndrome, toxic epidermal necrolysis.
  * Other irAEs: Severe infusion reactions, pancreatitis, uveitis, demyelination, autoimmune neuropathy (including facial and abducens nerve paresis), Guillain-Barré syndrome, myasthenia gravis, myasthenic syndrome, aseptic meningitis, encephalitis, gastritis, sarcoidosis, duodenitis, myositis, myocarditis, and rhabdomyolysis, Vogt-Koyanagi-Harada syndrome, hypoparathyroidism, cystitis noninfective; and
  * Other treatment-related AEs.
Severity (grade) of the following types of treatment-related AEs in the overall study population | Up to 157 weeks
  * Select irAEs: Immune-related pneumonitis, immune-related colitis, immune-related hepatitis, immune-related nephritis and renal dysfunction, immune-related endocrinopathies (hyperthyroidism, hypothyroidism, adrenal insufficiency, hypophysitis, diabetes mellitus and diabetic ketoacidosis), and immune-related skin adverse reactions (rash, Stevens-Johnson syndrome, toxic epidermal necrolysis.
  * Other irAEs: Severe infusion reactions, pancreatitis, uveitis, demyelination, autoimmune neuropathy (including facial and abducens nerve paresis), Guillain-Barré syndrome, myasthenia gravis, myasthenic syndrome, aseptic meningitis, encephalitis, gastritis, sarcoidosis, duodenitis, myositis, myocarditis, and rhabdomyolysis, Vogt-Koyanagi-Harada syndrome, hypoparathyroidism, cystitis noninfective; and
  * Other treatment-related AEs.
Seriousness of the following types of treatment-related AEs in the overall study population | Up to 157 weeks
  * Select irAEs: Immune-related pneumonitis, immune-related colitis, immune-related hepatitis, immune-related nephritis and renal dysfunction, immune-related endocrinopathies (hyperthyroidism, hypothyroidism, adrenal insufficiency, hypophysitis, diabetes mellitus and diabetic ketoacidosis), and immune-related skin adverse reactions (rash, Stevens-Johnson syndrome, toxic epidermal necrolysis.
  * Other irAEs: Severe infusion reactions, pancreatitis, uveitis, demyelination, autoimmune neuropathy (including facial and abducens nerve paresis), Guillain-Barré syndrome, myasthenia gravis, myasthenic syndrome, aseptic meningitis, encephalitis, gastritis, sarcoidosis, duodenitis, myositis, myocarditis, and rhabdomyolysis, Vogt-Koyanagi-Harada syndrome, hypoparathyroidism, cystitis noninfective; and
  * Other treatment-related AEs.
Outcome of the following types of treatment-related AEs in the overall study population | Up to 157 weeks
  * Select irAEs: Immune-related pneumonitis, immune-related colitis, immune-related hepatitis, immune-related nephritis and renal dysfunction, immune-related endocrinopathies (hyperthyroidism, hypothyroidism, adrenal insufficiency, hypophysitis, diabetes mellitus and diabetic ketoacidosis), and immune-related skin adverse reactions (rash, Stevens-Johnson syndrome, toxic epidermal necrolysis.
  * Other irAEs: Severe infusion reactions, pancreatitis, uveitis, demyelination, autoimmune neuropathy (including facial and abducens nerve paresis), Guillain-Barré syndrome, myasthenia gravis, myasthenic syndrome, aseptic meningitis, encephalitis, gastritis, sarcoidosis, duodenitis, myositis, myocarditis, and rhabdomyolysis, Vogt-Koyanagi-Harada syndrome, hypoparathyroidism, cystitis noninfective; and
  * Other treatment-related AEs.
Action taken with study treatment of the following types of treatment-related AEs in the overall study population | Up to 157 weeks
  * Select irAEs: Immune-related pneumonitis, immune-related colitis, immune-related hepatitis, immune-related nephritis and renal dysfunction, immune-related endocrinopathies (hyperthyroidism, hypothyroidism, adrenal insufficiency, hypophysitis, diabetes mellitus and diabetic ketoacidosis), and immune-related skin adverse reactions (rash, Stevens-Johnson syndrome, toxic epidermal necrolysis.
  * Other irAEs: Severe infusion reactions, pancreatitis, uveitis, demyelination, autoimmune neuropathy (including facial and abducens nerve paresis), Guillain-Barré syndrome, myasthenia gravis, myasthenic syndrome, aseptic meningitis, encephalitis, gastritis, sarcoidosis, duodenitis, myositis, myocarditis, and rhabdomyolysis, Vogt-Koyanagi-Harada syndrome, hypoparathyroidism, cystitis noninfective; and
  * Other treatment-related AEs.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Athens, Greece

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm